CLINICAL TRIAL: NCT05319821
Title: Increasing Physical Activity in Rural Pennsylvanians: PCP Participants
Brief Title: PA Moves Trial - PCP Participants
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Kathryn Schmitz, Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: STUDY22110036; R01CA268017 (NIH)
Record Dates: First submitted 2022-03-10; First posted 2022-04-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Behavior; Physical Activity
MeSH Terms: conditions — Behavior; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Intervention (Active Comparator): PCP participants in the practice cohort or the intervention group will receive the ECHO46 intervention via real-time, interactive videoconferencing through Zoom sessions held once weekly for 4 weeks (4 sessions total) at regularly scheduled times convenient to providers. Session topics will focus on training PCP participants to assess, advise, and refer patients to be more physically active, as well as provide evidence-based strategies they can use to supplement and sustain their communication efforts.
  Interventions: Behavioral: Receive ECHO training
- Delayed Intervention (Active Comparator): PCP participants will be offered the intervention in year 5.
  Interventions: Behavioral: Offered ECHO training in year 5

INTERVENTIONS:
Behavioral: Receive ECHO training — Active Intervention
  Arms: Active Intervention
Behavioral: Offered ECHO training in year 5 — Delayed Intervention
  Arms: Delayed Intervention

SUMMARY:
The purpose of this voluntary research study is to determine the impact of an ECHO intervention on the likelihood that rural primary care providers (PCP) will refer their physically inactive patients to be more active.

DETAILED DESCRIPTION:
People living in rural areas are diagnosed and die from cancer at higher rates than people living in cities. Physical activity has been shown to decrease the risk and occurrence of a variety of cancers, including bladder, breast, colon, endometrial, gastric, kidney, and prostate cancers. Being inactive can cause over 10% of breast and colon cancer cases.

Compared to people living in cities, people living in rural areas tend to be less physically active. They're also more likely to be overweight/obese or have diabetes. Adults who are overweight, obese, or diabetic often have changes in the way their bodies deal with insulin, glucose metabolism, and inflammation. Physical activity is thought to reduce the risk of cancer by improving these issues over time.

PCPs and their staff can identify a patient's need for more physical activity, but may not have the time or resources to give advice or assistance. We have set up a telephone-based physical activity coaching program, called the MoveLine, to give inactive patients advice and assistance in becoming more physically active.

The purpose of this study is to determine if an ECHO intervention will impact the likelihood that PCPs will refer patients to the MoveLine for physical activity coaching.

Approximately 32-48 providers will take part in this research study.

ELIGIBILITY:
Inclusion Criteria:

1. Primary care providers or adjunct faculty from Primary Health Network (PHN) or UPMC clinics serving rural populations
2. Must be able to provide and understand informed consent

Exclusion Criteria:

1. Primary care providers or adjunct faculty NOT from PHN or UPMC clinics

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2022-09-21 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Likelihood of patient referral | Through study completion, an average of 5 years
  Percentage of participating primary care providers referring their patients to a community-level, telephone-based physical activity counseling service assessed through the EMR of their participating patients

SECONDARY OUTCOMES:
PAQ-M | Baseline intervention group vs. Baseline delayed intervention group
  The 11-question Morgenstern Physical Activity Questionnaire (PAQ-M) is a self-report of physical activity resulting from recreational activities, exercises, home or work activities, and chores.
Estimated average metabolic equivalents expended daily | 1 week at baseline
  Daily metabolic equivalents collected using an accelerometer from Actigraph
Estimated metabolic equivalents expended weekly | 1 week at baseline
  Weekly metabolic equivalents collected using an accelerometer from Actigraph, expressed in hours/week
Time in Sleep | 1 week at baseline
  Weekly time in sleep collected using an accelerometer from Actigraph
Sedentary Time | 1 week at baseline
  Weekly sedentary time collected using an accelerometer from Actigraph
Low physical activity | 1 week at baseline
  Weekly low physical activity collected using an accelerometer from Actigraph
Moderate physical activity | 1 week at baseline
  Weekly moderate physical activity collected using an accelerometer from Actigraph
Vigorous physical activity | 1 week at baseline
  Weekly vigorous physical activity collected using an accelerometer from Actigraph

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Schmitz, PhD, Principal Investigator — University of Pittsburgh
Locations (2):
- United States (2):
  - Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - UPMC, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No